CLINICAL TRIAL: NCT04359108
Title: Environmental Localization Mapping and Guidance for Visual Prosthesis Users
Acronym: SLAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Carnegie Mellon University (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00228932; 1R01EY029741-01A1 (NIH)
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Retinitis Pigmentosa; Visual Impairment; Visual Prosthesis
Keywords: Retinal Prosthesis; Argus II
MeSH Terms: conditions — Retinitis Pigmentosa; Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Evaluation of normally sighted participants using a simulated visual prosthesis (Experimental): All normally sighted participants will be assigned to this arm of the study. This study group will perform all experiments using a virtual reality headset (Oculus Go) to simulate the limited vision of a retinal prosthesis system. This study group will include all interventions, including those that both match and exceed the visual performance of the Argus II system.
  Interventions: Device: Navigation system mode: Argus Vision; Device: Navigation system mode: Depth Vision; Device: Navigation system mode: Depth Vision with Haptic / Audio; Device: Navigation system mode: Haptic / Audio; Device: Navigation system mode: High Field-of-View Depth Vision; Device: Distance test vision mode: Low Resolution / Low Field-of-View; Device: Distance test vision mode: Low Resolution / High Field-of-View; Device: Distance test vision mode: High Resolution / Low Field-of-View; Device: Distance test vision mode: High Resolution / High Field-of-View
- Evaluation of blind participants using the Argus II retinal prosthesis (Experimental): All blind participants who have been implanted with the Argus II Retinal Prosthesis System will be assigned to this arm of the study. This study group will be limited to performing a subset of the interventions including only those that do not exceed the visual performance of the Argus II system.
  Interventions: Device: Navigation system mode: Argus Vision; Device: Navigation system mode: Depth Vision; Device: Navigation system mode: Depth Vision with Haptic / Audio; Device: Navigation system mode: Haptic / Audio; Device: Distance test vision mode: Low Resolution / Low Field-of-View

INTERVENTIONS:
Device: Navigation system mode: Argus Vision — This intervention uses the navigational aid with the output sensory modalities configured as follows:
  * Vision: Argus mode
  * Haptics: none
  * Audio: none Since this mode only provides the standard Argus vision, it is equivalent to using the base Argus II system without the navigational aid.
Device: Navigation system mode: Depth Vision — This intervention uses the navigational aid with the output sensory modalities configured as follows:
  * Vision: Depth mode (at Argus II resolution and field-of-view)
  * Haptics: none
  * Audio: none
Device: Navigation system mode: Depth Vision with Haptic / Audio — This intervention uses the navigational aid with the output sensory modalities configured as follows:
  * Vision: Depth mode (at Argus II resolution and field-of-view)
  * Haptics: yes
  * Audio: yes
Device: Navigation system mode: Haptic / Audio — This intervention uses the navigational aid with the output sensory modalities configured as follows:
  * Vision: none
  * Haptics: yes
  * Audio: yes Since this mode does not provide any visual feedback, it is equivalent to using navigational aid completely blind without a visual prosthesis.
Device: Navigation system mode: High Field-of-View Depth Vision — This intervention uses the navigational aid with the output sensory modalities configured as follows:
  * Vision: High Field-of-View Depth mode (at twice the Argus II resolution and field-of-view along each dimension)
  * Haptics: none
  * Audio: none
  Arms: Evaluation of normally sighted participants using a simulated visual prosthesis
Device: Distance test vision mode: Low Resolution / Low Field-of-View — This intervention performs the relative distance to two obstacles test with the user's vision output configured as follows:
  * Resolution: Low
  * Field-of-View: Low
Device: Distance test vision mode: Low Resolution / High Field-of-View — This intervention performs the relative distance to two obstacles test with the user's vision output configured as follows:
  * Resolution: Low
  * Field-of-View: High
  Arms: Evaluation of normally sighted participants using a simulated visual prosthesis
Device: Distance test vision mode: High Resolution / Low Field-of-View — This intervention performs the relative distance to two obstacles test with the user's vision output configured as follows:
  * Resolution: High
  * Field-of-View: Low
  Arms: Evaluation of normally sighted participants using a simulated visual prosthesis
Device: Distance test vision mode: High Resolution / High Field-of-View — This intervention performs the relative distance to two obstacles test with the user's vision output configured as follows:
  * Resolution: High
  * Field-of-View: High
  Arms: Evaluation of normally sighted participants using a simulated visual prosthesis

SUMMARY:
This study is driven by the hypothesis that independent navigation by blind users of visual prosthetic devices can be greatly aided by use of an autonomous navigational aid that provides information about the environment and guidance for navigation through multimodal sensory cues. For this study, the investigators developed a navigation system that uses on-board sensing to map the user's environment and compute navigable paths to desired destinations in real-time. Information regarding obstacles and directional guidance is communicated to the user via a combination of sensory modalities including limited vision (through the user's visual prosthesis), haptic, and audio cues. This study evaluates how effectively this navigational aid improves prosthetic vision users' ability to perform navigational tasks. The participants for this study include both retinal prosthesis users of the Argus II Retinal Prosthesis System (Argus II) and normally sighted individuals who use a virtual reality headset to simulate the limited vision of the Argus II system.

DETAILED DESCRIPTION:
About 1.3 million Americans aged 40 and older are legally blind, a majority because of diseases with onset later in life, such as glaucoma and age-related macular degeneration. Second Sight Medical Products (SSMP) has developed the world's first FDA approved retinal implant, Argus II, intended to restore some functional vision for people suffering from retinitis pigmentosa (RP).

In this era of smart devices, generic navigation technology, such as GPS mapping apps for smartphones, can provide directions to help guide a blind user from point A to point B. However, these navigational aids do little to enable blind users to form an egocentric understanding of the surroundings, are not suited to navigation indoors, and do nothing to assist in avoiding obstacles to mobility. The Argus II, on the other hand, provides blind users with a limited visual representation of the users surroundings that improves users' ability to orient themselves and traverse obstacles, yet lacks features for high-level navigation and semantic interpretation of the surroundings. The proposed study aims to address these limitations of the Argus II through a synergy of state-of-the-art simultaneous localization and mapping (SLAM) and scene recognition technologies.

This study is driven by the hypothesis that independent navigation by blind users of visual prosthetic devices can be greatly aided by use of an autonomous navigational aid that provides information about the environment and guidance for navigation through multimodal sensory cues. The investigators developed a navigation system that uses on-board sensing and SLAM-based algorithms to continuously construct a map of the user's environment and locate the user within that map in real-time. On-board path planning algorithms compute optimal navigation routes to reach desired destinations based on the constructed map. The system then communicates obstacle locations and navigational cues to the user while navigating via a combination of sensory modalities. The participants for this study include blind Argus II users, who use their retinal implant for vision, and normally sighted individuals, who use a virtual reality headset to simulate the limited vision of a retinal prosthesis.

The sensory modalities used by the navigational aid to communicate information back to the user include:

* Limited vision is provided via the user's visual prosthesis, with the Argus II retinal implant supporting an image size of 10 x 6 pixels spanning approximately 18 x 11 degrees field-of-view. Images sent to the visual implant are derived from video frames provided by forward-facing cameras integrated within headgear worn by the user. Three forms of vision feedback are evaluated in this study including: 1) the standard vision output of the Argus II (which uses texture-based processing including difference-of-Gaussian and contrast enhancement filters), 2) an enhanced depth-based vision mode that uses the depth sensing capabilities of the navigational aid to highlight above-ground obstacles, and 3) a high field of view depth-based vision mode that doubles the pixel size and field of view of the visual feedback in each dimension. The depth-vision modes display only above-ground obstacles with increasing brightness relative to decreasing distance from the user; the ground and obstacles beyond a threshold distance are not displayed in order to declutter the visual scene. The high field-of-view depth-vision mode is only utilized by normally sighted participants, as this mode exceeds the vision capabilities of the Argus II implant.
* Haptic cues indicate the direction in which the user should advance in order to follow the path computed by the navigational aid to reach a target destination. The haptic cues are generated by vibrators situated at five positions located left-to-right along the users forehead, which are built into user-worn headgear. The five vibration points indicate for the user to turn in directions: "far left", "slight left", "straight ahead", "slight right", and "far right".
* Audio cues provide an audible alert when the user approaches an obstacle within 1.5 feet and provide verbal updates on the remaining distance to reach the destination along the path computed by the navigational aid.

This study compares participants' performance in completing navigation tasks using five different modes and combinations of the foregoing sensory modalities as follows: 1) Argus vision, 2) depth vision, 3) depth vision with haptic and audio, 4) haptic and audio (without vision), and 5) high field-of-view depth vision.

The navigation tasks performed by the participants using these modalities include navigating through a dense obstacle field and navigating between rooms within an indoor facility that requires successful traversal of non-trivial paths.

In addition, a third experiment evaluates the effect of resolution and field-of-view of the retinal implant upon participants' ability to visually discern relative distances to different obstacles based on optical flow patterns induced by the participant's motion when approaching obstacles situated at different distances ahead of the user. For this experiment, the following four vision settings are evaluated: 1) low resolution / low field-of-view, 2) low resolution / high field-of-view, 3) high resolution / low field-of-view, and 4) high resolution / high field-of-view. The "low" settings correspond to the values of the Argus II system, whereas the "high" settings corresponding to a doubling of the "low" values along each dimension. For Argus user participants, only the low resolution / low field-of-view setting is evaluated since the Argus II retinal implant is incapable of supporting the higher vision settings.

ELIGIBILITY:
Criteria for inclusion of normally sighted individuals:

* Subject speaks English;
* Subjects must be an adult (at least 18 years of age);
* Subject has the cognitive and communication ability to participate in the study (i.e., follow spoken directions, perform tests, and give feedback);
* Subject is willing to conduct psychophysics testing up to 4-6 hours per day of testing on 3-5 consecutive days;
* Subject has visual acuity of 20/40 or better (corrected);
* Subject is capable of understanding participant information materials and giving written informed consent.
* Subject is able to walk unassisted

Criteria for inclusion of Argus II users:

The inclusion criteria for the study are the following:

* Subject is at least 25 years of age;
* Subject has been implanted with the Argus II system;
* Subject's eye has healed from surgery and the surgeon has cleared the subject for programming;
* Subject has the cognitive and communication ability to participate in the study (i.e., follow spoken directions, perform tests, and give feedback);
* Subject is willing to conduct psychophysics testing up to 4-6 hours per day of testing on 3-5 consecutive days;
* Subject is capable of understanding patient information materials and giving written informed consent;
* Subject is able to walk unassisted.

Exclusion criteria for all subjects is the following:

* Subject is unwilling or unable to travel to testing facility for at least 3 days of testing within a one-week timeframe;
* Subject does not speak English;
* Subject has language or hearing impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth Billings, Ph.D., Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Medicine - Wilmer Eye Institute, Baltimore, Maryland
  - Johns Hopkins Applied Physics Laboratory, Laurel, Maryland

IPD SHARING:
Plan to Share IPD: No
Results from this study will be disseminated through conference presentations and peer-reviewed publications. However, IPD will not be shared outside the study team.

REFERENCES:
- [Derived] Christie B, Norena Acosta N, Sadeghi R, Kartha A, Ewulum C, Caspi A, Tenore FV, Dagnelie G, Klatzky RL, Billings SD. Autonomous multisensory enhancement of a visual neuroprosthesis for navigation: Technical proof-of-concept with simulated prosthetic vision and single-subject case study of a visual prosthesis user. J Neural Eng. 2026 Jan 26. doi: 10.1088/1741-2552/ae3d67. Online ahead of print. PMID 41587489

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For blind participants, 6 individuals who had previously received the Argus II retinal implant were recruited.
  For sighted participants, 20 individuals with normal vision were recruited from staff members of the Johns Hopkins University Applied Physics Laboratory.
Period: Overall Study
Arm/Group | Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis | Evaluation of Blind Participants Using the Argus II Retinal Prosthesis
Started | 20 | 6
Completed | 19 | 1
Not Completed | 1 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Unable or too feeble to walk independently | 0 | 2
Not completed — Argus II system stopped functioning | 0 | 1
Not completed — Died of natural causes unrelated to the study before study ended | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis | Evaluation of Blind Participants Using the Argus II Retinal Prosthesis | Total
Number analyzed (Participants) | 20 | 6 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 2 | 21
  >=65 years | 1 | 4 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 14 | 4 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 6 | 18
  Unknown or Not Reported | 8 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 9 | 6 | 15
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 5 | 0 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 6 | 26
Vision Impairment [Count of Participants; unit: Participants]
  Normal Vision | 20 | 0 | 20
  Blind having Argus II Implant | 0 | 6 | 6

OUTCOME MEASURES:

1. Primary Outcome: Duration of Time to Complete Navigational Tasks as Assessed by the Mean Duration of Travel in Seconds Normalized by the Nominal Path Distance in Meters
Description: Participants will be asked to complete the navigation tasks of crossing an obstacle field approximately 6 meters in length and navigating to a target destination located about 20 - 30 meters away. The normalized duration of time to complete each navigation task will be measured in seconds. To account for variability in the path distances of different trials, the measured time will be normalized by a reference (nominal) path distance in meters associated with the configuration of each trial. The mean normalized time across all trials will be computed for each intervention.
Time Frame: Up to 7 minutes for each navigation task, on Day 1 or Day 2
Population: Participants who completed the task are reported
Measure: Mean (Standard Error); unit: seconds/meter
Arm/Group | Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis | Evaluation of Blind Participants Using the Argus II Retinal Prosthesis
Number analyzed (Participants) | 20 | 1
seconds/meter
  Obstacle Field Test: Argus Vision | 14.54 (1.03) | 14.09 (2.19)
  Obstacle Field Test: Depth Vision | 10.46 (0.93) | 14.60 (2.17)
  Obstacle Field Test: Depth Vision + Haptic/Audio | 9.38 (0.80) | 14.05 (1.31)
  Obstacle Field Test: Haptic/Audio | 9.72 (0.83) | 9.13 (1.29)
  Obstacle Field Test: High Field-of-View Depth Vision | 7.54 (0.68) | NA (NA) — Prosthetic implant for Argus II users does not support wide field-of-view vision of this intervention.
  Navigate to Destination Test: Argus Vision | 9.32 (0.94) | NA (NA) — Intended destination was not successfully reached in any trials for this task and intervention, therefore statistics cannot be computed.
  Navigate to Destination Test: Depth Vision | 8.68 (0.81) | 5.11 (NA) — Intended destination was successfully reached in only 1 trial for this task and intervention, therefore standard error cannot be computed.
  Navigate to Destination Test: Depth Vision + Haptic/Audio | 7.05 (0.44) | 7.95 (1.70)
  Navigate to Destination Test: Haptic/Audio | 7.05 (0.49) | 9.31 (1.75)
  Navigate to Destination Test: High Field-of-View Depth Vision | 6.37 (0.59) | NA (NA) — Prosthetic implant for Argus II users does not support wide field-of-view vision of this intervention.
Statistical Analysis 1: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; Navigate to Destination Test - Significance of Navigation Mode: test for null hypothesis of equivalent performance among all navigation system modes; Test type: Other; p = 0.02, ANOVA
Statistical Analysis 2: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; Navigate to Destination Test - Argus Vision vs. Depth Vision: test for null hypothesis of equivalent performance; Test type: Other; p = 0.22, t-test, 2 sided
Statistical Analysis 3: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; Navigate to Destination Test - Depth Vision vs. Depth Vision + Haptic/Audio: test for null hypothesis of equivalent performance; Test type: Other; p = 0.017, t-test, 2 sided
Statistical Analysis 4: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; Navigate to Destination Test - Haptic/Audio vs. Depth Vision + Haptic/Audio: test for null hypothesis of equivalent performance; Test type: Other; p = 0.98, t-test, 2 sided
Statistical Analysis 5: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; Navigate to Destination Test - Depth Vision vs. High Field-of-View Depth Vision: test for null hypothesis of equivalent performance; Test type: Other; p = 0.014, t-test, 2 sided
Statistical Analysis 6: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; Obstacle Avoidance Test - Significance of Navigation Mode: test for null hypothesis of equivalent performance among all navigation system modes; Test type: Other; p < 0.001, ANOVA
Statistical Analysis 7: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; Obstacle Avoidance Test - Argus Vision vs. Depth Vision: test for null hypothesis of equivalent performance; Test type: Other; p < 0.01, t-test, 2 sided
Statistical Analysis 8: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; Obstacle Avoidance Test - Depth Vision vs. Depth Vision + Haptic/Audio: test for null hypothesis of equivalent performance; Test type: Other; p = 0.156, t-test, 2 sided
Statistical Analysis 9: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; Obstacle Avoidance Test - Haptic/Audio vs. Depth Vision + Haptic/Audio: test for null hypothesis of equivalent performance; Test type: Other; p = 0.541, t-test, 2 sided
Statistical Analysis 10: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; Obstacle Avoidance Test - Depth Vision vs. High Field-of-View Depth Vision: test for null hypothesis of equivalent performance; Test type: Other; p < 0.01, t-test, 2 sided
Statistical Analysis 11: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; Obstacle Avoidance Test - Argus Vision: test for null hypothesis that the single Argus participant in this arm has performance that lies in-distribution with performance statistics computed for the normally sighted subjects arm of the study; Test type: Other; Test Method: Z-Score comparison of the performance of the single Argus participant to the performance distribution of normally sighted subjects. Significance threshold: |Z| = 2.8 for p = 0.05, 2-tailed (reject null hypothesis above threshold) Result: Z-Score = -0.10
Statistical Analysis 12: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; Obstacle Avoidance Test - Depth Vision: test for null hypothesis that the single Argus participant in this arm has performance that lies in-distribution with performance statistics computed for the normally sighted subjects arm of the study; Test type: Other; Test Method: Z-Score comparison of the performance of the single Argus participant to the performance distribution of normally sighted subjects. Significance threshold: |Z| = 2.8 for p = 0.05, 2-tailed (reject null hypothesis above threshold) Result: Z-Score = 1.00
Statistical Analysis 13: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; Obstacle Avoidance Test - Depth Vision + Haptic/Audio: test for null hypothesis that the single Argus participant in this arm has performance that lies in-distribution with performance statistics computed for the normally sighted subjects arm of the study; Test type: Other; Test Method: Z-Score comparison of the performance of the single Argus participant to the performance distribution of normally sighted subjects. Significance threshold: |Z| = 2.8 for p = 0.05, 2-tailed (reject null hypothesis above threshold) Result: Z-Score = 0.88
Statistical Analysis 14: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; Obstacle Avoidance Test - Haptic/Audio: test for null hypothesis that the single Argus participant in this arm has performance that lies in-distribution with performance statistics computed for the normally sighted subjects arm of the study; Test type: Other; Test Method: Z-Score comparison of the performance of the single Argus participant to the performance distribution of normally sighted subjects. Significance threshold: |Z| = 2.8 for p = 0.05, 2-tailed (reject null hypothesis above threshold) Result: Z-Score = -1.6
Statistical Analysis 15: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; Navigate to Destination Test - Argus Vision: test for null hypothesis that the single Argus participant in this arm has performance that lies in-distribution with performance statistics computed for the normally sighted subjects arm of the study; Test type: Other; Test Method: Z-Score comparison of the performance of the single Argus participant to the performance distribution of normally sighted subjects. Significance threshold: |Z| = 2.8 for p = 0.05, 2-tailed (reject null hypothesis above threshold) Result: Z-Score = N/A * * N/A for Argus Vision test because subject did not successfully reach intended destination for any trial using this mode
Statistical Analysis 16: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; Navigate to Destination Test - Depth Vision: test for null hypothesis that the single Argus participant in this arm has performance that lies in-distribution with performance statistics computed for the normally sighted subjects arm of the study; Test type: Other; Test Method: Z-Score comparison of the performance of the single Argus participant to the performance distribution of normally sighted subjects. Significance threshold: |Z| = 2.8 for p = 0.05, 2-tailed (reject null hypothesis above threshold) Result: Z-Score = -1.10
Statistical Analysis 17: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; Navigate to Destination Test - Depth Vision + Haptic/Audio: test for null hypothesis that the single Argus participant in this arm has performance that lies in-distribution with performance statistics computed for the normally sighted subjects arm of the study; Test type: Other; Test Method: Z-Score comparison of the performance of the single Argus participant to the performance distribution of normally sighted subjects. Significance threshold: |Z| = 2.8 for p = 0.05, 2-tailed (reject null hypothesis above threshold) Result: Z-Score = 0.45
Statistical Analysis 18: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; Navigate to Destination Test - Haptic/Audio: test for null hypothesis that the single Argus participant in this arm has performance that lies in-distribution with performance statistics computed for the normally sighted subjects arm of the study; Test type: Other; Test Method: Z-Score comparison of the performance of the single Argus participant to the performance distribution of normally sighted subjects. Significance threshold: |Z| = 2.8 for p = 0.05, 2-tailed (reject null hypothesis above threshold) Result: Z-Score = 1.02

2. Primary Outcome: Distance Traversed to Complete Navigational Tasks as Assessed by the Mean Distance Traveled in Meters Normalized by the Nominal Path Distance in Meters
Description: Participants will be asked to complete the navigation tasks of crossing an obstacle field approximately 6 meters in length and navigating to a target destination located about 20 - 30 meters away. The normalized distance traversed to complete each navigation task will be measured. To account for variability in the path distances of different trials, the measured distance will be normalized by a reference (nominal) path distance in meters associated with the configuration of each trial. The mean normalized distance across all trials will be computed for each intervention.
Time Frame: Up to 7 minutes for each navigation task, on Day 1 or Day 2
Population: Participants who completed the task are reported
Measure: Mean (Standard Error); unit: meters/meter
Arm/Group | Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis | Evaluation of Blind Participants Using the Argus II Retinal Prosthesis
Number analyzed (Participants) | 20 | 1
meters/meter
  Obstacle Field Test: Argus Vision | 1.598 (0.045) | 1.543 (0.048)
  Obstacle Field Test: Depth Vision | 1.305 (0.027) | 1.427 (0.126)
  Obstacle Field Test: Depth Vision + Haptic/Audio | 1.227 (0.018) | 1.537 (0.125)
  Obstacle Field Test: Haptic/Audio | 1.230 (0.026) | 1.300 (0.095)
  Obstacle Field Test: High Field-of-View Depth Vision | 1.217 (0.025) | NA (NA) — Prosthetic implant for Argus II users does not support wide field-of-view vision of this intervention.
  Navigate to Destination Test: Argus Vision | 1.236 (0.095) | NA (NA) — Intended destination was not successfully reached in any trial for this task and intervention, therefore statistics cannot be computed.
  Navigate to Destination Test: Depth Vision | 1.315 (0.075) | 1.1 (NA) — Intended destination was successfully reached in only 1 trials for this task and intervention, therefore standard error cannot be computed.
  Navigate to Destination Test: Depth Vision + Haptic/Audio | 1.130 (0.034) | 1.505 (0.245)
  Navigate to Destination Test: Haptic/Audio | 1.138 (0.035) | 1.735 (0.205)
  Navigate to Destination Test: High Field-of-View Depth Vision | 1.196 (0.072) | NA (NA) — Prosthetic implant for Argus II users does not support wide field-of-view vision of this intervention.
Statistical Analysis 1: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.30, ANOVA
Statistical Analysis 2: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; [analysis description as in outcome 1, analysis 6]; Test type: Other; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; Obstacle Avoidance Test - Argus Vision vs. Depth Vision: test for null hypothesis of equivalent performance; Test type: Other; p < 0.01, t-test, 2 sided
Statistical Analysis 4: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; [analysis description as in outcome 1, analysis 8]; Test type: Other; p = 0.01, t-test, 2 sided
Statistical Analysis 5: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; [analysis description as in outcome 1, analysis 9]; Test type: Other; p = 0.93, t-test, 2 sided
Statistical Analysis 6: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; [analysis description as in outcome 1, analysis 10]; Test type: Other; p < 0.01, t-test, 2 sided
Statistical Analysis 7: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; [analysis description as in outcome 1, analysis 11]; Test type: Other; Test Method: Z-Score comparison of the performance of the single Argus participant to the performance distribution of normally sighted subjects. Significance threshold: |Z| = 2.8 for p = 0.05, 2-tailed (reject null hypothesis above threshold) Result: Z-Score = -0.27
Statistical Analysis 8: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; [analysis description as in outcome 1, analysis 12]; Test type: Other; [other analysis details as in outcome 1, analysis 12]
Statistical Analysis 9: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; [analysis description as in outcome 1, analysis 13]; Test type: Other; Test Method: Z-Score comparison of the performance of the single Argus participant to the performance distribution of normally sighted subjects. Significance threshold: |Z| = 2.8 for p = 0.05, 2-tailed (reject null hypothesis above threshold) Result: Z-Score = 2.75
Statistical Analysis 10: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; [analysis description as in outcome 1, analysis 14]; Test type: Other; Test Method: Z-Score comparison of the performance of the single Argus participant to the performance distribution of normally sighted subjects. Significance threshold: |Z| = 2.8 for p = 0.05, 2-tailed (reject null hypothesis above threshold) Result: Z-Score = 0.60
Statistical Analysis 11: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; [analysis description as in outcome 1, analysis 15]; Test type: Other; Test Method: Z-Score comparison of the performance of the single Argus participant to the performance distribution of normally sighted subjects. Significance threshold: |Z| = 2.8 for p = 0.05, 2-tailed (reject null hypothesis above threshold) Result: Z-Score = N/A* * N/A for Argus Vision test because subject did not successfully reach intended destination for any trial using this mode
Statistical Analysis 12: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; [analysis description as in outcome 1, analysis 16]; Test type: Other; Test Method: Z-Score comparison of the performance of the single Argus participant to the performance distribution of normally sighted subjects. Significance threshold: |Z| = 2.8 for p = 0.05, 2-tailed (reject null hypothesis above threshold) Result: Z-Score = -0.72
Statistical Analysis 13: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; [analysis description as in outcome 1, analysis 15]; Test type: Other; Test Method: Z-Score comparison of the performance of the single Argus participant to the performance distribution of normally sighted subjects. Significance threshold: |Z| = 2.8 for p = 0.05, 2-tailed (reject null hypothesis above threshold) Result: Z-Score = 2.47
Statistical Analysis 14: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; [analysis description as in outcome 1, analysis 15]; Test type: Other; Test Method: Z-Score comparison of the performance of the single Argus participant to the performance distribution of normally sighted subjects. Significance threshold: |Z| = 2.8 for p = 0.05, 2-tailed (reject null hypothesis above threshold) Result: Z-Score = 3.81

3. Primary Outcome: Obstacle Avoidance While Completing Navigational Tasks as Assessed by the Mean Number of Contacts With Obstacles Normalized by the Nominal Path Distance in Meters
Description: Participants will be asked to complete the navigation tasks of crossing an obstacle field approximately 6 meters in length and navigating to a target destination located about 20 - 30 meters away. The number of contacts with obstacles encountered while completing each navigation task will be measured. To account for variability in the path distances of different trials, the number of contacts will be normalized by a reference (nominal) path distance in meters associated with the configuration of each trial. The mean normalized number of contacts with obstacles across all trials will be computed for each intervention.
Time Frame: Up to 7 minutes for each navigation task, on Day 1 or Day 2
Population: Participants who completed the task are reported
Measure: Mean (Standard Error); unit: number of contacts / meter
Arm/Group | Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis | Evaluation of Blind Participants Using the Argus II Retinal Prosthesis
Number analyzed (Participants) | 20 | 1
number of contacts / meter
  Obstacle Field Test: Argus Vision | 0.737 (0.060) | 0.523 (0.101)
  Obstacle Field Test: Depth Vision | 0.224 (0.039) | 0.465 (0.058)
  Obstacle Field Test: Depth Vision + Haptic/Audio | 0.201 (0.025) | 0.175 (0.101)
  Obstacle Field Test: Haptic/Audio | 0.250 (0.035) | 0.116 (0.116)
  Obstacle Field Test: High Field-of-View Depth Vision | 0.090 (0.029) | NA (NA) — Prosthetic implant for Argus II users does not support wide field-of-view vision of this intervention.
  Navigate to Destination Test: Argus Vision | 0.407 (0.057) | NA (NA) — Intended destination was not successfully reached in any trials for this task and intervention, therefore statistics cannot be computed.
  Navigate to Destination Test: Depth Vision | 0.257 (0.055) | 0.297 (NA) — Intended destination was successfully reached in only 1 trial for this task and intervention, therefore standard error cannot be computed.
  Navigate to Destination Test: Depth Vision + Haptic/Audio | 0.130 (0.017) | 0.054 (0.013)
  Navigate to Destination Test: Haptic/Audio | 0.151 (0.016) | 0.061 (0.006)
  Navigate to Destination Test: High Field-of-View Depth Vision | 0.162 (0.035) | NA (NA) — Prosthetic implant for Argus II users does not support wide field-of-view vision of this intervention.
Statistical Analysis 1: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.001, ANOVA; navigation system mode and test block as factors
Statistical Analysis 2: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; Navigate to Destination Test - Argus Vision vs. Depth Vision: test for null hypothesis of equivalent performance; Test type: Other; p < 0.01, t-test, 2 sided; within-participant, 2 sided t-test
Statistical Analysis 3: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; [analysis description as in outcome 1, analysis 3]; Test type: Other; p = 0.037, t-test, 2 sided — within-participant, 2 sided t-test
Statistical Analysis 4: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; [analysis description as in outcome 1, analysis 4]; Test type: Other; p = 0.34, t-test, 2 sided; within-participant, 2 sided t-test
Statistical Analysis 5: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; [analysis description as in outcome 1, analysis 5]; Test type: Other; p = 0.10, t-test, 2 sided; within-participant, 2 sided t-test
Statistical Analysis 6: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; [analysis description as in outcome 1, analysis 6]; Test type: Other; p < 0.001, ANOVA
Statistical Analysis 7: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; Obstacle Avoidance Test - Argus Vision vs. Depth Vision: test for null hypothesis of equivalent performance; Test type: Other; p < 0.01, t-test, 2 sided
Statistical Analysis 8: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; [analysis description as in outcome 1, analysis 8]; Test type: Other; p = 0.67, t-test, 2 sided
Statistical Analysis 9: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; [analysis description as in outcome 1, analysis 9]; Test type: Other; p = 0.23, t-test, 2 sided
Statistical Analysis 10: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; [analysis description as in outcome 1, analysis 10]; Test type: Other; p < 0.01, t-test, 2 sided
Statistical Analysis 11: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; [analysis description as in outcome 1, analysis 11]; Test type: Other; Test Method: Z-Score comparison of the performance of the single Argus participant to the performance distribution of normally sighted subjects. Significance threshold: |Z| = 2.8 for p = 0.05, 2-tailed (reject null hypothesis above threshold) Result: Z-Score = -0.79
Statistical Analysis 12: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; [analysis description as in outcome 1, analysis 12]; Test type: Other; Test Method: Z-Score comparison of the performance of the single Argus participant to the performance distribution of normally sighted subjects. Significance threshold: |Z| = 2.8 for p = 0.05, 2-tailed (reject null hypothesis above threshold) Result: Z-Score = 1.38
Statistical Analysis 13: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; [analysis description as in outcome 1, analysis 13]; Test type: Other; Test Method: Z-Score comparison of the performance of the single Argus participant to the performance distribution of normally sighted subjects. Significance threshold: |Z| = 2.8 for p = 0.05, 2-tailed (reject null hypothesis above threshold) Result: Z-Score = 2.24
Statistical Analysis 14: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; [analysis description as in outcome 1, analysis 14]; Test type: Other; Test Method: Z-Score comparison of the performance of the single Argus participant to the performance distribution of normally sighted subjects. Significance threshold: |Z| = 2.8 for p = 0.05, 2-tailed (reject null hypothesis above threshold) Result: Z-Score = -0.85
Statistical Analysis 15: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; [analysis description as in outcome 1, analysis 15]; Test type: Other; [other analysis details as in outcome 2, analysis 11]
Statistical Analysis 16: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; [analysis description as in outcome 1, analysis 16]; Test type: Other; Test Method: Z-Score comparison of the performance of the single Argus participant to the performance distribution of normally sighted subjects. Significance threshold: |Z| = 2.8 for p = 0.05, 2-tailed (reject null hypothesis above threshold) Result: Z-Score = 0.18
Statistical Analysis 17: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; [analysis description as in outcome 1, analysis 17]; Test type: Other; Test Method: Z-Score comparison of the performance of the single Argus participant to the performance distribution of normally sighted subjects. Significance threshold: |Z| = 2.8 for p = 0.05, 2-tailed (reject null hypothesis above threshold) Result: Z-Score = -0.97
Statistical Analysis 18: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis vs Evaluation of Blind Participants Using the Argus II Retinal Prosthesis; [analysis description as in outcome 1, analysis 15]; Test type: Other; Test Method: Z-Score comparison of the performance of the single Argus participant to the performance distribution of normally sighted subjects. Significance threshold: |Z| = 2.8 for p = 0.05, 2-tailed (reject null hypothesis above threshold) Result: Z-Score = -1.23

4. Primary Outcome: Success in Completing Navigational Tasks as Assessed by the Mean Percentage of Trials Where Participants Successfully Reached the Intended Destination
Description: Participants will be asked to navigate to a target destination located about 20 - 30 meters away. We will measure success rate as the mean number of trials for which each participants successfully reached the intended destination divided by the total number of trials performed by that participant for each intervention.
Time Frame: Up to 7 minutes for each navigation task, on Day 1 or Day 2
Population: Participants who completed the task are reported
Measure: Mean (Standard Error); unit: percentage of trials
Arm/Group | Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis | Evaluation of Blind Participants Using the Argus II Retinal Prosthesis
Number analyzed (Participants) | 20 | 1
percentage of trials
  Argus Vision | 50.0 (8.9) | 0 (NA) — Standard error cannot be measured due to having only 1 measured value from 1 participant.
  Depth Vision | 65.7 (8.6) | 50 (NA) — Standard error cannot be measured due to having only 1 measured value from 1 participant.
  Depth Vision + Haptic / Audio | 97.5 (2.5) | 100 (NA) — Standard error cannot be measured due to having only 1 measured value from 1 participant.
  Haptic / Audio | 92.5 (4.1) | 100 (NA) — Standard error cannot be measured due to having only 1 measured value from 1 participant.
  High Field of View Depth Vision | 72.5 (7.7) | 100 (NA) — Standard error cannot be measured due to having only 1 measured value from 1 participant.
Statistical Analysis 1: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.001, ANOVA; Single-factor test on navigation system mode
Statistical Analysis 2: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; Navigate to Destination Test - Argus Vision vs. Depth Vision: test for null hypothesis of equivalent performance; Test type: Other; p = 0.17, t-test, 2 sided
Statistical Analysis 3: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; [analysis description as in outcome 1, analysis 3]; Test type: Other; p < 0.01, t-test, 2 sided
Statistical Analysis 4: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; [analysis description as in outcome 1, analysis 4]; Test type: Other; p = 0.33, t-test, 2 sided
Statistical Analysis 5: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; [analysis description as in outcome 1, analysis 5]; Test type: Other; p < 0.01, t-test, 2 sided

5. Primary Outcome: Accuracy of Relative Distance Judgments as Assessed by the Percentage of Correct Responses
Description: Participants will be presented with two physical objects and asked to identify which of the objects is the nearer one after walking a controlled distance down a centerline oriented between the objects. We will measure accuracy as the percentage of correct responses (the total number of correct responses divided by the total number of trials times 100).
Time Frame: Up to 60 seconds for each discrimination task, on Day 1 or Day 2
Population: Participants who completed the task are reported
Measure: Mean (Standard Error); unit: percentage of correct responses
Arm/Group | Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis | Evaluation of Blind Participants Using the Argus II Retinal Prosthesis
Number analyzed (Participants) | 10 | 1
percentage of correct responses
  Low Resolution / Low Field-of-View | 62 (3.4) | 83 (NA) — Standard error cannot be measured due to having only 1 measured value from 1 participant.
  Low Resolution / High Field-of-View | 72.2 (3.9) | NA (NA) — Prosthetic implant for Argus II users does not support the high field-of-view vision of this mode.
  High Resolution / Low Field-of-View | 67.8 (4.4) | NA (NA) — Prosthetic implant for Argus II users does not support the high resolution vision of this mode.
  High Resolution / High Field-of-View | 75.6 (2.9) | NA (NA) — Prosthetic implant for Argus II users does not support the high resolution and high field-of-view vision of this mode.
Statistical Analysis 1: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; Significance of Resolution: test for null hypothesis of equivalent performance between low and high resolution vision modes; Test type: Other; p = 0.023, ANOVA; 2X2 within-participant test with factors of resolution and field-of-view
Statistical Analysis 2: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; Significance of Resolution: test for null hypothesis of equivalent performance between low and high field-of-view vision modes; Test type: Other; p = 0.039, ANOVA; 2X2 within-participant test with factors of resolution and field-of-view
Statistical Analysis 3: Comparison: Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis; Significance of Interaction between Resolution and Field-of-View: test for null hypothesis of no interaction; Test type: Other; p = .801, ANOVA; 2x2 within-participant test with factors of resolution and field-of-view

ADVERSE EVENTS:
Time Frame: Up to 2 days
Arm/Group | Evaluation of Normally Sighted Participants Using a Simulated Visual Prosthesis | Evaluation of Blind Participants Using the Argus II Retinal Prosthesis
All-Cause Mortality (participants affected / at risk) | 0/20 | 2/6
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/6
Other Adverse Events (participants affected / at risk) | 0/20 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT04359108/Prot_SAP_000.pdf